CLINICAL TRIAL: NCT05627791
Title: Effects of Vaginal Oxytocin Gel on Vaginal Cytologic Parameters in Postmenopausal Woman: A Randomized Placebo-controlled Trial
Brief Title: Effects of Vaginal Oxytocin Gel on Vaginal Cytologic Parameters in Postmenopausal Woman
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unable to recuit participant number in time.
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 65065
Record Dates: First submitted 2022-11-09; First posted 2022-11-28 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Vaginal Atrophy; Oxytocin Gel; Postmenopausal Women; Vaginal Maturation Index
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin gel (Experimental): Oxytocin gel 400IU per 1 ml (on HPMC 4,000 cps base gel), applied at vaginal canal 1 ml per day for 8 weeks
  Interventions: Drug: Oxytocin
- Placebo gel (Placebo Comparator): Placebo gel (HPMC 4,000 cps base gel) , applied at vaginal canal 1 ml per day for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin vaginal gel that have oxytocin 400IU/1ml of gel, base gel contained HPMC 4,000 cps, 5% propylene glycol USP, 0.08% methylparaben, sterile water for irrigation and 0.02% propylparaben then adjusted pH by Lactic acid and sodium hydroxide keep pH 3.5-4.0
  Other Names: Oxytocin vaginal gel
  Arms: Oxytocin gel
Drug: Placebo — Placebo gel that have base gel contained HPMC 4,000 cps, 5% propylene glycol USP, 0.08% methylparaben, sterile water for irrigation and 0.02% propylparaben then adjusted pH by Lactic acid and sodium hydroxide keep pH 3.5-4.0 without oxytocin
  Arms: Placebo gel

SUMMARY:
Vulvovaginal atrophy affects around 90% of postmenopausal women who may present with symptoms such as dryness, irritation, itching, burning, and dyspareunia that negatively affect the quality of life. Topical estrogen is recommended for the treatment of vulvovaginal atrophy in postmenopausal women and the FDA approved it. But it may increase the risk of breast and endometrial cancer. The oxytocin hormone also promotes positive social behavior, stress regulation, and female sexual arousal. Many previous studies show that topical oxytocin is useful for reducing vaginal atrophy in postmenopausal women.

DETAILED DESCRIPTION:
Random and conducted on 56 postmenopausal women who meet the inclusion criteria and excluded participants that have exclusion criteria. All women provided written informed consent before data collection.

1. st Visit: The vagina was assessed regarding infection and any abnormal discharge. The participants were evaluated vaginal signs of vaginal atrophy by per vaginal examination and assessed vaginal health index score. The subjective symptoms were assessed by The most bothersome score. The vaginal pH was tested with a Nitrazine paper. The vaginal swab was done and the specimen was sent for a cytological test - vaginal maturation index evaluation (VMI). The participants were separated into two groups 1. Oxytocin gel group and 2. Placebo gel group then applied gel 1 ml. (400IU of oxytocin in oxytocin gel) per day for 8 weeks consecutively. The subjective symptoms were assessed at 2 and 4 weeks by phone.
2. nd Visit: The participants were assessed the same as 1st visit that recorded vaginal health index score, subjective symptoms, vaginal pH, and vaginal maturation index evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Thai menopausal women aged between 50-70 years who visit Rajavithi gynecology OPD with informed consent with good communication in the Thai language.

Exclusion Criteria:

* Have acute vulvovaginitis (vaginal swab for wet smear and KOH)
* Patients who have used hormonal replacement therapy within 12 months
* Patients with a history of smoking
* Patients who have used vaginal lubricant or moisturizer
* Patients with an allergic history of oxytocin or gel components
* Morbid obesity BMI > 30 kg/m2
* Patients who have used vitamin E supplement
* Patients who unable to perform per vaginal examination

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Comparison of vaginal cytology test for vaginal maturation index measurement | Change from baseline VMI at 8 weeks
  VMI = 0.2 × % parabasal cells+0.6 × % intermediate cells+1.0 × % superficial cells score below 52 mean significant vulvovaginal atrophy

SECONDARY OUTCOMES:
Comparison of vaginal health index; scoring from vaginal examination | Change from baseline vaginal health index score at 8 weeks
  Score 5-25, below 15 mean significant vulvovaginal atrophy from physical examination
Comparison of subjective symptoms by The most bothersome symptoms score | Change from baseline subjective symptom score at 2 weeks
  score from 0-4, 0 = absent, 4 = severe symptom
Comparison of subjective symptoms by The most bothersome symptoms score | Change from baseline subjective symptom score at 4 weeks
  score from 0-4, 0 = absent, 4 = severe symptom
Comparison of subjective symptoms by The most bothersome symptoms score | Change from baseline subjective symptom score at 8 weeks
  score from 0-4, 0 = absent, 4 = severe symptom
Comparison of vaginal pH between two group | Vaginal pH at 8 weeks
  pH from Nitrazine paper test
Comparison of adverse events between two group | adverse events within 8 weeks
  present of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zohrabi I, Abedi P, Ansari S, Maraghi E, Shakiba Maram N, Houshmand G. The effect of oxytocin vaginal gel on vaginal atrophy in postmenopausal women: a randomized controlled trial. BMC Womens Health. 2020 May 19;20(1):108. doi: 10.1186/s12905-020-00935-5. PMID 32429977
- [Background] Alvisi S, Gava G, Orsili I, Giacomelli G, Baldassarre M, Seracchioli R, Meriggiola MC. Vaginal Health in Menopausal Women. Medicina (Kaunas). 2019 Sep 20;55(10):615. doi: 10.3390/medicina55100615. PMID 31547180
- [Background] Gandhi J, Chen A, Dagur G, Suh Y, Smith N, Cali B, Khan SA. Genitourinary syndrome of menopause: an overview of clinical manifestations, pathophysiology, etiology, evaluation, and management. Am J Obstet Gynecol. 2016 Dec;215(6):704-711. doi: 10.1016/j.ajog.2016.07.045. Epub 2016 Jul 26. PMID 27472999
- [Background] Jonasson AF, Edwall L, Uvnas-Moberg K. Topical oxytocin reverses vaginal atrophy in postmenopausal women: a double-blind randomized pilot study. Menopause Int. 2011 Dec;17(4):120-5. doi: 10.1258/mi.2011.011030. Epub 2011 Nov 25. PMID 22120944
- [Background] Fianu Jonasson A, Bixo M, Sundstrom Poromaa I, Astrom M. Safety and Efficacy of an Oxytocin Gel and an Equivalent Gel but Without Hormonal Ingredients (Vagivital(R) Gel) in Postmenopausal Women with Symptoms of Vulvovaginal Atrophy: A Randomized, Double-Blind Controlled Study. Med Devices (Auckl). 2020 Oct 5;13:339-347. doi: 10.2147/MDER.S265824. eCollection 2020. PMID 33116956
- [Background] Kallak TK, Uvnas-Moberg K. Oxytocin stimulates cell proliferation in vaginal cell line Vk2E6E7. Post Reprod Health. 2017 Mar;23(1):6-12. doi: 10.1177/2053369117693148. Epub 2017 Mar 8. PMID 28381099
- [Background] Hess R, Austin RM, Dillon S, Chang CC, Ness RB. Vaginal maturation index self-sample collection in mid-life women: acceptability and correlation with physician-collected samples. Menopause. 2008 Jul-Aug;15(4 Pt 1):726-9. doi: 10.1097/gme.0b013e31816c5541. PMID 18427354
- [Background] Torky HA, Taha A, Marie H, El-Desouky E, Raslan O, Moussa AA, Ahmad AM, Abo-Louz A, Zaki S, Fares T, Eesa A. Role of topical oxytocin in improving vaginal atrophy in postmenopausal women: a randomized, controlled trial. Climacteric. 2018 Apr;21(2):174-178. doi: 10.1080/13697137.2017.1421924. Epub 2018 Jan 19. PMID 29347848
- [Background] Al-Saqi SH, Uvnas-Moberg K, Jonasson AF. Intravaginally applied oxytocin improves post-menopausal vaginal atrophy. Post Reprod Health. 2015 Sep;21(3):88-97. doi: 10.1177/2053369115577328. Epub 2015 May 19. PMID 25995333